CLINICAL TRIAL: NCT07203963
Title: Additional Effects of Niel Asher Technique Along With Sleeper Stretch on Posterior Capsule in Patients With Adhesive Capsulitis.
Brief Title: Additional Effects of Niel-asher Technique on Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maria Barket
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Adhesive Capsulitis
Keywords: Niel-Asher Technique (NAT); Sleeper stretch; trigger points
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niel-Asher Technique+ sleeper stretch+ Conventional PT (Other): Niel-Asher Technique
  Interventions: Other: Niel-Asher Technique + sleeper stretch
- sleeper stretch + Conventional Treatment (Other): Sleeper stretch+ Conventional
  Interventions: Other: sleeper stretch + Conventional Treatment

INTERVENTIONS:
Other: Niel-Asher Technique + sleeper stretch — Niel-Asher Technique, Manual Soft Tissue releaser, Neuro-muscular release technique for adhesive capsulitis ( This manual technique will be applied for 3 days a week for 4 weeks).Sleeper stretch will be applied passively by investigator, pressure of the stretch will be held for 30 seconds (repeated twice with 30 seconds break for 3 days a week) Conventional PT including 1: shoulder anteroposterior, posteroanterior and inferior glides ( 3 times a week for 4 week) 2: active and active assisted ROM exercises of shoulder joint (frequency: 1 set of 10 repetitions twice a day). 3: Shoulder Isometric exercises, Codman's exercises and pulley and finger ladder exercises (frequency: 1 set of 10 repetitions twice a day), 4: trigger points will be released by applying ischemic pressure (90 seconds) on trigger points found in rotator cuff muscles.
  Arms: Niel-Asher Technique+ sleeper stretch+ Conventional PT
Other: sleeper stretch + Conventional Treatment — Sleeper stretch will be applied passively by investigator, pressure of the stretch will be held for 30 seconds (repeated twice with 30 seconds break for 3 days a week). Conventional PT including 1: shoulder anteroposterior, posteroanterior and inferior glides ( 3 times a week for 4 week) 2: active and active assisted ROM exercises of shoulder joint (frequency: 1 set of 10 repetitions twice a day). 3: Shoulder Isometric exercises, Codman's exercises and pulley and finger ladder exercises (frequency: 1 set of 10 repetitions twice a day) 4: ischemic compression (90seconds hold) on trigger points found in rotator cuff muscles
  Arms: sleeper stretch + Conventional Treatment

SUMMARY:
The aim of this randomized controlled trial is to find the additional effects of Niel-Asher technique along with sleeper stretch and conventional physical therapy on pain, shoulder ranges of motion and functional disability in patients with Adhesive capsulitis

DETAILED DESCRIPTION:
Frozen shoulder is a musculoskeletal disorder and it is a painful shoulder condition, it is also known as adhesive capsulitis. This condition is usually caused by progressive fibrosis and contracture of glenohumeral joint capsule and it cause pain and stiffness in glenohumeral joint. In patients with adhesive capsulitis there is significant reduction of both active and passive ROMs. Adhesive capsulitis is more common in females than in males with the age range from 40-60 years. Most affected ROM in patient with adhesive capsulitis is external rotation but internal rotation and other range of motions of shoulder are also affected. Frozen shoulder is prevalent in 2-3% of general population, with variations across countries and regions. There are three stages of adhesive capsulitis. Patient in early stages usually present with inflammation which progressively changes into fibrotic changes. Its diagnosis is usually made on the basis of history and physical examination.

Shoulder joint capsule has different segments and each segment has some effect on shoulder ROMs in all directions. Thickness of joint capsule is primary restraint that cause reduction in ROMs in frozen shoulder patient. Fibrosis of glenohumeral joint capsule often cause effusion of long head of bicep brachi. Risk factor for adhesive capsulitis includes female gender specifically age greater than 45 and diabetes, Dupuytren contracture, immobilization of the shoulder, complex regional pain syndrome. Individuals with higher BMI with hyperlipidemia are at higher risk for adhesive capsulitis. A study on subjects with chronic non traumatic shoulder pain (n=72) showed high prevalence of MTrPs in all subjects; highest prevalence being in infraspinatus (78%) followed by upper trapezius (58%), middle trapezius (43%), deltoid and teres minor.

Niel-Asher technique mainly based on the principle of body's natural healing mechanisms. It targets adherent structures to release fibrosis. It also stimulates specific neural pathways by activating mechanoreceptors and helps CNS to enhance pain reduction and functional improvement. This technique remodels the shoulder capsule by relieving soft tissue adhesions. It also decreases nociceptive sensitivity, improves circulation that leads to pain relief and restoration of range of motion of shoulder joint. This technique employed deep stroking massage and compression of trigger points in five steps on major muscles such as rotator cuff muscles/ teres minor, Infraspinatus and deltoid muscle.

Sleeper stretch technique isolates the soft tissue restraints in the posterior shoulder to correct mobility and flexibility deficit. Sleeper stretch targets infraspinatus and teres minor muscles and improve shoulder ROMs and internal rotation by decreasing stiffness of the posterior capsule and muscle tendon tension.

This study aims to find the additional effect of Niel-Asher technique along with sleeper stretch and conventional therapy (which include exercise therapy and ischemic compression to release trigger points )on minimizing pain, improving shoulder ranges of motion and functional activities in individuals affected by Adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Both Genders: Male and Female
* Patient falls under diagnostic criteria for adhesive capsulitis which is Painful and limited active and passive glenohumeral ROM in capsular pattern (external rotation> abduction> internal rotation)
* Patient diagnosed with adhesive capsulitis by orthopedic or general physician
* Patient with phase two and three of adhesive capsulitis based on duration of symptoms
* Patients of adhesive capsulitis with presence of trigger points in rotator cuff muscles and deltoid muscle (trigger points present in at least 1 or 2 of these muscles) based on simon and travell's criteria of trigger points diagnosis.

Exclusion Criteria:

* Spinal Injuries and any other co- morbidity
* Any surgery, infection, trauma, pregnancy, fracture and fall
* Patient with intra articular steroidal therapy with in last 6 months
* Patient unwilling to comply follow up schedule
* Patient involvement in another intervention study
* Malignancy
* Patient with thyroid disorders and RA and Glenohumeral OA
* History of previous surgery or manipulation under anesthesia of affected shoulder
* Patient with duration of symptoms of less than three months

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue scale VAS | 4 weeks
  It is a pain rating scale. The findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain. Patient will be asked to verbally report the pain score
Shoulder pain and disability Index (SPADI) | 4 weeks
  The shoulder pain and disability index (SPADI) was developed to measure Current shoulder pain and disability, it is widely used valid and reliable tool. The SPADI contains 13 items that assess two domains, a 5-item subscale that measures pain and 8-item subscale that measures disability.
Goniometer | 4 weeks
  A goniometer will be used to measure the range of motion (ROM) of the Shoulder joint. Goniometer is an instrument that measures the available range of motion at a joint

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Shafi International Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No